CLINICAL TRIAL: NCT06773468
Title: Evaluating Knowledge Mobilization for Stress Management in University Students
Brief Title: Evaluating Knowledge Mobilization Vehicles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Nancy Heath, Distinguished James McGill Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-11-006; SSHRC 430-2022-00172 (Other Grant/Funding Number: Social Sciences and Humanities Research Council)
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Stress; Coping; Digital Intervention; University Students
Keywords: stress; coping; digital intervention; self-directed; online resource; university students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Workshop (Experimental): 30-minute online stress management workshop providing psychoeducation and strategy practice with links to strategies shared at the end
  Interventions: Behavioral: stress management
- Video (Experimental): a short 10-minute stress management video providing psychoeducation and strategy practice with links to strategies shared at the end
  Interventions: Behavioral: stress management
- Infographic (Experimental): a brief 3-page stress management interactive infographic (i.e., with psychoeducation and embedded links for strategy practice)
  Interventions: Behavioral: stress management
- Inactive control (No Intervention): Waitlist inactive control that will receive all stress management materials at the end of the study

INTERVENTIONS:
Behavioral: stress management — These different stress management modalities have been developed to ensure equivalent content across: (a) psychoeducation and strategy introduction; and (b) skills-based practice of strategies. Stress management strategies touched on 4 main areas which included (a) pause/break; (b) positive awareness; (c) kindness to self; and (d) social support.
  Arms: Infographic; Video; Workshop

SUMMARY:
The present study examined the comparative effectiveness of self-directed (video, infographic) vs. non-self directed (workshop) modalities of online stress management resources and an inactive control condition in terms of their effectiveness and acceptability for university students.

DETAILED DESCRIPTION:
University students have been reporting high levels of stress, which have been found to negatively impact their academic performance and overall well-being. Given these elevated levels of stress, a large number of students report using unhealthy coping behaviours such as alcohol and drug use or risky sexual behaviours to cope with daily stressors. High levels of stress can be harmful to students' quality of life and well-being (both physical and mental), as well as elevated stress over an extended period can hinder academic performance. To address the overwhelming demands for wellness services, online approaches to delivering stress management and well-being supports are being used on campuses as supplemental means of promoting student stress management, coping capacity, and well-being.

Growing research on the barriers associated with help-seeking and changes due to the pandemic have spurred a shift from in-person supports to online self-directed modalities. Evidence from research measuring the acceptability of digital mental health interventions in university students suggests that students rate these interventions with moderate to high acceptability, but students report concerns around the use of certain digital modalities such as privacy, credibility, and lack of guidance on how to get started and use the interventions. Research has demonstrated how these types of online support can be effective at enhancing university student well-being and decreasing stress. For example, an umbrella review of systematic reviews and meta-analyses to synthesize the literature on digital mental health interventions in higher education found that most interventions were effective at decreasing depression symptoms, anxiety, and stress in this context. Specifically, skills-training and cognitive behavioral therapy (CBT)-based interventions were found to be effective. However, it is important to highlight that the authors found that the effectiveness depended on the modality or delivery format of the intervention. Although there is evidence for their individual effectiveness when compared to inactive control groups, it is crucial to have a better theoretical understanding of their relative effectiveness to one another to make research-informed decisions in selecting instructional approaches to support students' coping capacity in higher education.

Therefore, the overarching objective of the current study is to investigate how stress management knowledge can be effectively put into action within the university context by comparing different modalities. The study seeks to investigate differences in response to self-directed vs. non self-directed approaches to sharing stress management knowledge with students against a control group, specifically in terms of acceptability and change over time on wellness outcomes while accounting for the role of strategy use frequency. Specifically, the first objective (1.1) was to compare and evaluate self-directed, non self-directed, and an inactive control group by assessing effectiveness as demonstrated in changes (pre/post/follow-up) on wellness outcomes (i.e., perceived stress, coping capacity, mindfulness, coping self-efficacy, and well-being), while (1.2) examining the role of strategy use frequency. The second objective (2) is to further examine specific differences between commonly used knowledge mobilization modalities for stress management strategies (workshop, video, infographic) and an inactive control group by assessing (2.1) acceptability (i.e., likelihood of use, satisfaction) and (2.2) effectiveness as demonstrated in changes (pre/post/follow-up) on the same wellness outcomes while (2.3) examining the role of strategy use frequency.

ELIGIBILITY:
Inclusion Criteria:

* Current university student

Exclusion Criteria:

-

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 313 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Stress | Week 0, 4, and 7
  The Perceived Stress Scale (PSS) is a widely used self-report measure of individuals' perception of stress. This measure contains 10 items in which participants indicate their experience of stress on a 5-point Likert scale (0 = never to 4 = very often). Items were adapted to reflect experiences during the past week and include statements such as "In the past week, how often have you felt difficulties were piling up so high that you could not overcome them?" Ratings were averaged across items such that higher scores represented greater perceived stress. The PSS has good reliability (Cronbach's α = .89), construct validity, and predictive validity with reports of psychological and physical symptoms.

SECONDARY OUTCOMES:
Change in Satisfaction | Week 4 and 7
  The Response to Training is a researcher-developed questionnaire assessing participants' satisfaction with the intervention content and delivery. The questions were delivered according to the three levels of Kirkpatrick's New World Model (Kirkpatrick & Kirkpatrick, 2016) as follows: (1) student viewers' response (i.e., satisfaction, engagement, relevance); (2) learning (i.e., knowledge, skills, attitude, confidence, commitment); (3) use of skills (i.e., willingness to use, frequency of use). All items are scored on a 6-point Likert-scales except for the strategy use item described below, where higher scores represent a better response to training. Sample items include "I would recommend the stress management resource to other university students" or "I am planning to use the strategies in the future..."
Change in coping capacity | Week 0, 4, and 7
  The Coping Index (CI; (Stallman, 2017), a 20-item measure of engagement with healthy and unhealthy coping strategies that are aligned with the health theory of coping framework (Stallman, 2020). The measure consists of items that list common healthy and unhealthy coping behaviours such as 'talk things over with family or friends', 'do relaxing activities', or 'have negative self-talk'. Participants are asked to indicate how often they engage in each behaviour listed when they feel stressed or distressed on a 4-point Likert scale (0 = I don't do this at all to 3 = I do this most of the time). This measure has been found to have satisfactory test-retest reliability with alpha = 0.71 (Stallman, 2019).
Change in mindfulness | Week 0, 4, and 7
  The Five Facets of Mindfulness Questionnaire short form (FFMQ-15; (Baer et al., 2006, 2008) which is a 15-item self-report measure consisting of five subscales each assessing a specific facet of dispositional mindfulness: acting with awareness, describing, observing, non-reactivity, and non-judgmental acceptance. Items include "I'm good at finding words to describe my feelings" and "When I have distressing thoughts or images, I am able just to notice them without reacting". Participants rate their responses on a 5-point Likert scale (1 = never or very rarely true to 5 = very often or always true). The FFMQ-15 has good internal consistency with Cronbach alphas ranging from .64 to .83, as well as convergent validity (Gu et al., 2016). Higher scores on the FFMQ-15 represent higher mindfulness.
Change in coping self-efficacy | Week 0, 4, and 7
  The Coping Self-Efficacy Scale (CSES; Chesney et al., 2006) which is a measure of one's confidence in effectively engaging in coping behaviors in the face of challenges. This measure contains 26 items in which participants indicate confidence in their coping strategies when it comes to handling challenges and stressors on an 11-point Likert scale (0 = cannot do at all to 10 = certain can do). The CSES states, "When things aren't going well for you, or when you're having problems, how confident or certain are you that you can do the following:" and include statements such as "find solutions to your most difficult problems" and "see things from the other person's point of view during a heated argument." Higher scores on the CSES represent higher coping-self efficacy.
Change in well-being | Week 0, 4, and 7
  The Warwick-Edinburg Mental Well-Being Scale (WEMWBS; Tennant et al., 2007), which is a measure of positive mental health and consists of 14 positively worded items. Participants are asked to rate statements such as "I've been feeling good about yourself" on a 5-point Likert scale according to their experience over the past 2 weeks (1= none of the time; 5= all of the time). The WEMWBS has demonstrated good internal consistency in student (α = .89) and general population samples (α = .91) and was found to be psychometrically robust in validation studies (Stewart-Brown et al., 2011; Tennant et al., 2007).

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Restricted by our ethics board approval.

REFERENCES:
- [Background] Harith S, Backhaus I, Mohbin N, Ngo HT, Khoo S. Effectiveness of digital mental health interventions for university students: an umbrella review. PeerJ. 2022 Mar 31;10:e13111. doi: 10.7717/peerj.13111. eCollection 2022. PMID 35382010
- [Background] Lattie EG, Adkins EC, Winquist N, Stiles-Shields C, Wafford QE, Graham AK. Digital Mental Health Interventions for Depression, Anxiety, and Enhancement of Psychological Well-Being Among College Students: Systematic Review. J Med Internet Res. 2019 Jul 22;21(7):e12869. doi: 10.2196/12869. PMID 31333198
- [Background] Bourdon JL, Moore AA, Long EC, Kendler KS, Dick DM. The relationship between on-campus service utilization and common mental health concerns in undergraduate college students. Psychol Serv. 2020 Feb;17(1):118-126. doi: 10.1037/ser0000296. Epub 2018 Oct 8. PMID 30299149
- [Background] LaMontagne LG, Doty JL, Diehl DC, Nesbit TS, Gage NA, Kumbkarni N, Leon SP. Acceptability, usage, and efficacy of mindfulness apps for college student mental health: A systematic review and meta-analysis of RCTs. J Affect Disord. 2024 Dec 15;367:951-971. doi: 10.1016/j.jad.2024.09.014. Epub 2024 Sep 10. PMID 39260578
- [Background] Harrer M, Adam SH, Baumeister H, Cuijpers P, Karyotaki E, Auerbach RP, Kessler RC, Bruffaerts R, Berking M, Ebert DD. Internet interventions for mental health in university students: A systematic review and meta-analysis. Int J Methods Psychiatr Res. 2019 Jun;28(2):e1759. doi: 10.1002/mpr.1759. Epub 2018 Dec 26. PMID 30585363
- [Background] Kern A, Hong V, Song J, Lipson SK, Eisenberg D. Mental health apps in a college setting: openness, usage, and attitudes. Mhealth. 2018 Jun 30;4:20. doi: 10.21037/mhealth.2018.06.01. eCollection 2018. PMID 30050916
- [Background] Frazier P, Gabriel A, Merians A, Lust K. Understanding stress as an impediment to academic performance. J Am Coll Health. 2019 Aug-Sep;67(6):562-570. doi: 10.1080/07448481.2018.1499649. Epub 2018 Oct 4. PMID 30285563
- [Background] Metzger IW, Blevins C, Calhoun CD, Ritchwood TD, Gilmore AK, Stewart R, Bountress KE. An examination of the impact of maladaptive coping on the association between stressor type and alcohol use in college. J Am Coll Health. 2017 Nov-Dec;65(8):534-541. doi: 10.1080/07448481.2017.1351445. Epub 2017 Jul 14. PMID 28708021